CLINICAL TRIAL: NCT07143396
Title: Evaluation of a Mind-Body Application in Combination With a Graded Movement Program for the Treatment of Chronic Pain
Brief Title: Evaluation of a Mind-Body Based Approach for Chronic Pain Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Fraser Valley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101806
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Migraine; Chronic Pain Syndrome
Keywords: mind-body; mobile application; chronic pain; guided movement; Somatic Education
MeSH Terms: conditions — Chronic Pain; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: All participants will be enrolled in the intervention arm: 6 weeks of engagement with a mind-body mobile application and virtual somatic education program. Results of the current study will be compared to two groups from the researcher's previous study, NCT05090683 (a usual care control group and a mobile app-only intervention group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-body mobile application and guided movement (Experimental): Participants are asked to engage (minimum 4x per week) with a user-guided mobile application (app) that employs mind-body techniques including expressive writing, meditation, cognitive behavioural therapy, and pain education. The app also includes access to podcasts that focus on pain counselling and pain education. Participants are also asked to follow (3x per week) an audio-guided somatic education program (light-intensity graded movement).
  Interventions: Behavioral: Mind-body mobile application and guided movement

INTERVENTIONS:
Behavioral: Mind-body mobile application and guided movement — Self-directed: The study team recommends daily use of the mobile app for 6 weeks, with a minimum of 4 times per week, and engagement with the somatic education program at least 3 times per week for 6 weeks. Frequency of app usage and somatic education engagement will be monitored via weekly surveys.

SUMMARY:
The investigators are evaluating the effects of a mind-body mobile application, in combination with a guided movement program, on the experience of chronic pain. Participants meeting the criteria for chronic/persistent pain (confirmed via self-report) will complete an online baseline questionnaire. Eligible participants will take part in an intervention that involves use of a 6-week free trial of a mind-body focused mobile application in combination with virtual asynchronous audio-guided somatic education sessions (gentle movement). External data from a usual care control arm and a mobile-app-only arm from a previous study by the same research team, National Clinical Trials (NCT) registry number NCT05090683, will be used for comparison with the current combined intervention. All participants will complete online surveys at the start of the study and after 6 weeks to measure pain intensity and interference (primary outcomes), mental health outcomes (depression, anxiety, stress), pain-related thoughts (pain catastrophizing), quality of life, and fear of movement (secondary outcomes). From weeks 2 to 6, participants will fill out weekly surveys to track how often they engage with each: the somatic education (gentle movement) program and the mobile app. Participants will also complete a follow-up survey at 12 weeks (6 weeks post-intervention conclusion).

DETAILED DESCRIPTION:
See protocol for more details. (submitted at time of registration)

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 19 to 75 years with chronic pain
* Chronic pain is defined as having non-malignant chronic or persistent pain for at least 6 months.
* Participants must experience pain at least half the days in the last 6 months.
* Pain can include bodily pain or head (migraine) pain
* Participants must have access to an electronic device
* Participants must be willing to engage in weekly somatic education activities

Exclusion Criteria:

* Individuals reporting a cognitive impairment that can interfere with completing questionnaires and using a mobile application.
* Individuals reporting substance use disorder (within the last 6 months).
* Individuals reporting any of the following medical conditions: metastatic cancer, rheumatoid arthritis, lupus, scleroderma, polymyositis.
* Individuals with previous experience with the mind-body app under study (Note: use of "Calm" or another meditation-only app is not an exclusion).
* Individuals with current regular (at least once a week) engagement with a somatic movement program (e.g., Feldenkrais, Hanna Somatics, Somatic Yoga, Tai Chi, Pilates)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory-short form (BPI-SF) Pain Severity | Baseline, 6 weeks.
  Measures self reported pain severity (over past 24 hours).
  BPI Pain Severity: single item scale within larger Brief Pain Inventory tool that asses pain "average" pain severity. Item scale ranges from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome (pain severity), lower scores indicate better outcome.
  Item range = (0,10).
Change in Brief Pain Inventory-short form (BPI-SF) Pain Interference | Baseline, 6 weeks.
  Item 9 on the BPI measures interference with daily living. There are 7 items (reflecting seven daily activities) and each is scored on 11-point scales from 0 = "does not interfere" to 10 = "completely interferes" for interference with activities of daily living. Pain interference score is calculated as an average of the 7 items, with a range from 0 to 10. Higher scores represent worse outcomes (higher interference).

SECONDARY OUTCOMES:
Change in Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity short form 3a | Baseline, 6 weeks, 12 weeks
  Measures self reported pain intensity over the past 7 days "on average" and "at its worst" along with an item to assess pain intensity "now". The three items are added together to produce a raw score which can be converted to a t-score.
  Each item uses 5-pt Likert scale from 1 = "had no pain" to 5 = "very severe".
  Raw scores range from 3 to 15. Higher scores indicate worse outcomes.
Change in Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference short form 8a | Baseline, 6 weeks, 12 weeks
  Measures self reported pain interference in daily activities (over 7 days). 8 items are added together for a raw score, which can then be converted to a t-score.
  Each item uses 5-pt Likert scale from 1 = "not at all" to 5 = "very much" (regarding pain interference).
  Raw scores range from 8 to 40. Higher scores indicate worse outcomes.
Change in Pain Catastrophizing Questionnaire (PCS) | Baseline, 6 and 12 weeks
  Measures thoughts and perceptions of pain, 13 items, scored using 5-pt Likert scale 0 = "not at all" to 4 = "all the time".
  Scores are the sum of all items. min score = 0; max score = 52. Higher scores indicate worse outcomes.
Change in Depression, Anxiety, and Stress Scale (DASS-21) | Baseline, 6 and 12 weeks
  Measures self reported emotional states, three subscales: depression, anxiety, stress (each 7 items) Items scored on 4-point Likert scale: 0 = "did not apply to me at all" to 3 = "applied to me very much or most of the time".
  Scores for each subscale are summed. Scores are then multiplied by 2 to calculate final score for each subscale.
  Scale ranges for each subscale is from 0 to 42 (after doubling of scores). Higher scores indicate worse outcomes.
Change in Quality of Life Short Form 12 (SF-12) Physical Component Score | Baseline, 6 and 12 weeks
  Measures self-reported impact of health on daily life. The SF-12 is a brief version of the SF-36 and contains 12 items measured using a variety of Likert scales and dichotomous yes/no scales, with each item response assigned a numerical weight.
  The Physical Component Score (PCS) is a summary score that is reported as a z-score. Scores are calculated using regression weights and constants that have been derived from a U.S. population.
  Each item response choice category is coded as an indicator variable (scored 1 / 0). Indicator variables are weighted using regression coefficients from the US population for the PCS. The weighted scores across all items are then summed and are added to a constant (regression intercept) to obtain a summary score. Score ranges 0 to 100. Normalized score such that component scales have a mean of 50 and standard deviation of 10 in the general population.
  Lower scores indicate worse outcomes. Higher scores indicate improved physical health.
Change in Quality of Life Short Form 12 (SF-12) Mental Component Score | Baseline, 6 and 12 weeks
  Measures self-reported impact of health on daily life. The SF-12 is a brief version of the SF-36 and contains 12 items measured using a variety of Likert scales and dichotomous yes/no scales, with each item response assigned a numerical weight.
  The Mental Component Score (MCS) is a summary score that is reported as a z-score. Scores are calculated using regression weights and constants that have been derived from a U.S. population.
  Each item response choice category is coded as an indicator variable (scored 1 / 0). Indicator variables are weighted using regression coefficients from the US population for the MCS. The weighted scores across all items are then summed and are added to a constant (regression intercept) to obtain a summary score. Score ranges 0 to 100. Normalized score such that component scales have a mean of 50 and standard deviation of 10 in the general population.
  Lower scores indicate worse outcomes. Higher scores indicate improved mental health.
Change in Tampa Scale of Kinesiophobia Questionnaire (TSK) | Baseline, 6 and 12 weeks
  Measured self-reported kinesiophobia assessing fear of movement or re-injury due to pain.
  Each item rated on a 4-point Likert scale: 1 = "strongly disagree" to 4 = "strongly agree." Total score range = (11, 44). Higher scores indicate greater fear of movement and worse outcomes.
Change in Brief Pain Inventory Pain Severity Composite Score | baseline, 6 weeks, 12 weeks
  A composite score derived from the average of four items that assesses at its "worst", "least", "average" over the past 24 hours, along with "now". Item scales range from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome, lower scores indicate better outcome.
  Item range = (0,10).
Change in Brief Pain Inventory Pain Severity (from baseline to 12 weeks) | baseline, 12 weeks
  Note: This is a secondary outcome (change from 0 to 6 weeks is a primary outcome).
  Measures self reported pain severity and pain interference (over past 24 hours).
  BPI Pain Severity: single item scale within larger Brief Pain Inventory tool that inquires about "average" pain severity over the past 24 hours. Item scale ranges from 0 to 10. 0 = "no pain", 10 = "pain as bad as you can imagine". Higher scores indicate worse outcome, lower scores indicate better outcome.
  Item range = (0,10).
Change in Brief Pain Inventory Interference (from baseline to 12 weeks) | baseline, 12 weeks
  Note: This is a secondary outcome (change from 0 to 6 weeks is a primary outcome).
  Measures self reported pain interference (over past 24 hours).
  BPI Pain Interference: Item 9 on BPI measures interference with daily living. There are 7 items embedded within and each is scored on 11-point scales from 0 = "does not interfere" to 10 = "completely interferes" for interference with activities of daily living. Pain interference score is calculated as an average of the 7 items, with a range from 0 to 10. Higher scores represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Thomson, PhD, Principal Investigator — University of the Fraser Valley
Locations (1):
- University of the Fraser Valley, Chilliwack, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roelofs J, Goubert L, Peters ML, Vlaeyen JW, Crombez G. The Tampa Scale for Kinesiophobia: further examination of psychometric properties in patients with chronic low back pain and fibromyalgia. Eur J Pain. 2004 Oct;8(5):495-502. doi: 10.1016/j.ejpain.2003.11.016. PMID 15324781
- [Background] Kean J, Monahan PO, Kroenke K, Wu J, Yu Z, Stump TE, Krebs EE. Comparative Responsiveness of the PROMIS Pain Interference Short Forms, Brief Pain Inventory, PEG, and SF-36 Bodily Pain Subscale. Med Care. 2016 Apr;54(4):414-21. doi: 10.1097/MLR.0000000000000497. PMID 26807536
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Devan H, Farmery D, Peebles L, Grainger R. Evaluation of Self-Management Support Functions in Apps for People With Persistent Pain: Systematic Review. JMIR Mhealth Uhealth. 2019 Feb 12;7(2):e13080. doi: 10.2196/13080. PMID 30747715
- [Background] Schopflocher D, Taenzer P, Jovey R. The prevalence of chronic pain in Canada. Pain Res Manag. 2011 Nov-Dec;16(6):445-50. doi: 10.1155/2011/876306. PMID 22184555
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Morone NE, Greco CM. Mind-body interventions for chronic pain in older adults: a structured review. Pain Med. 2007 May-Jun;8(4):359-75. doi: 10.1111/j.1526-4637.2007.00312.x. PMID 17610459
- [Background] Pfeifer AC, Uddin R, Schroder-Pfeifer P, Holl F, Swoboda W, Schiltenwolf M. Mobile Application-Based Interventions for Chronic Pain Patients: A Systematic Review and Meta-Analysis of Effectiveness. J Clin Med. 2020 Nov 5;9(11):3557. doi: 10.3390/jcm9113557. PMID 33167300
- [Background] Ashar YK, Gordon A, Schubiner H, Uipi C, Knight K, Anderson Z, Carlisle J, Polisky L, Geuter S, Flood TF, Kragel PA, Dimidjian S, Lumley MA, Wager TD. Effect of Pain Reprocessing Therapy vs Placebo and Usual Care for Patients With Chronic Back Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jan 1;79(1):13-23. doi: 10.1001/jamapsychiatry.2021.2669. PMID 34586357
- [Background] Thomson CJ, Pahl H, Giles LV. Randomized controlled trial investigating the effectiveness of a multimodal mobile application for the treatment of chronic pain. Can J Pain. 2024 Aug 19;8(1):2352399. doi: 10.1080/24740527.2024.2352399. eCollection 2024. PMID 39175941

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT07143396/Prot_SAP_000.pdf